CLINICAL TRIAL: NCT00998413
Title: Secondary Prevention of Asthma in Overweight/Obese Children by a Combined Dietary-behavioural-physical Activity Intervention
Brief Title: Weight-reduction Intervention in Asthmatic Children With Overweight/Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: The Netherlands Asthma Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEC 09-2-088; NAF 3.4.09.002 (Other Grant/Funding Number: Dutch Asthma Foundation)
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Asthma; Overweight; Obesity
Keywords: asthma; overweight; obesity; children
MeSH Terms: conditions — Asthma; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifaceted intervention (Experimental): Multifaceted intervention:physical exercise, nutrition, and behavioural intervention.
  Interventions: Behavioral: Multifaceted intervention
- Control (No Intervention): standard usual care

INTERVENTIONS:
Behavioral: Multifaceted intervention — multifaceted family-based, physical exercise, nutrition, and behavioural intervention study for 18 month, in children aged 6-16 years with asthma and overweight/obesity.
  Other Names: MIKADO
  Arms: Multifaceted intervention

SUMMARY:
The purpose of this study is to determine the efficacy of a multifactorial intervention with weight reduction, behavioural therapy, and physical exercise on the severity and control of asthma in obese children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-16 years
* BMI in the overweight/obesity range according to data of Cole et al.
* Asthma diagnosis

Exclusion Criteria:

* Children with a normal weight according to data of Cole et al.
* Children without any provable asthmatic complaints
* Congenital malformations of the airways or other chronic lung diseases like cystic fibrosis (CF)
* Mental retardation or syndromes
* Heart disease

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2010-01; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in the first second (FEV1 %) predicted value | 2 years

SECONDARY OUTCOMES:
Airway inflammation | 2 years
Symptom-free days, exacerbations | 2 years
Need for beta-2 agonists/anti-inflammatory medication | 2 years
Weight, height, body mass index (BMI) | 2 years
Levels of serum adipokines | 2 years
aerobic capacity | 2 years
  VO2max measured with an maximal ergometry test

CONTACTS AND LOCATIONS:
Overall Officials: Edward Dompeling, PhD, MD, Principal Investigator — Maastricht University Medical Centre; Kim van de Kant, MSc, Study Chair — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Willeboordse M, van de Kant KDG, Tan FE, Mulkens S, Schellings J, Crijns Y, Ploeg Lv, van Schayck CP, Dompeling E. A Multifactorial Weight Reduction Programme for Children with Overweight and Asthma: A Randomized Controlled Trial. PLoS One. 2016 Jun 13;11(6):e0157158. doi: 10.1371/journal.pone.0157158. eCollection 2016. PMID 27294869
- [Derived] Willeboordse M, van de Kant KD, de Laat MN, van Schayck OC, Mulkens S, Dompeling E. Multifactorial intervention for children with asthma and overweight (Mikado): study design of a randomised controlled trial. BMC Public Health. 2013 May 21;13:494. doi: 10.1186/1471-2458-13-494. PMID 23692648